CLINICAL TRIAL: NCT05257070
Title: The Clinical Validation of a Dried Blood Spot Method for Vancomycin and Creatinine
Acronym: ADVANCED
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B.C.M. (Brenda) de Winter, Assistant Professor, Erasmus Medical Center
Other Study IDs: NL79269.078.21
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Vancomycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: fingerprick — In addition to the standard venous samples, dried blood spot samples trough a fingerprick will be collected.
  Other Names: dried blood spot sampling

SUMMARY:
A widely used antibiotic is vancomycin. To ensure adequate exposure to vancomycin, drug doses are adjusted based on whole-blood concentration measurements, a practice known as therapeutic drug monitoring (TDM). The need for TDM of vancomycin is well established, as described in several national and international guidelines, for dose-optimization in order to achieve successful treatment and to prevent toxicity and reduce microbial resistance. A sampling method for TDM that has become more popular over the recent years is dried blood spotting (DBS). DBS is a design of blood sampling consisting of positioning a drop of capillary blood, preferably taken from the finger, on filter paper. Unlike venous blood sampling (the current gold standard for TDM of vancomycin), DBS seems to have advantages for the patient. The finger prick is less invasive than venipuncture. DBS also enables patients to perform one or multiple finger prick(s) themselves, with the possibility to sample at multiple time points. Due to the fact that vancomycin is nephrotoxic, it would be very efficient and convenient to measure creatinine in the same dried blood spot as the vancomycin. This study is a clinical validation study to validate the DBS assay for vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical patients
* Aged 18 and over
* Able to understand written information and able to give informed consent
* Treated with vancomycin
* Able and willing to undergo a finger prick for dried blood spot sampling
* Able and willing to fill in a questionnaire

Exclusion Criteria:

* Unable to draw blood samples for study purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults receiving intravenous vancomycin
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
To clinically validate the DBS method for vancomycin and creatinine in comparison to venipuncture vancomycin and creatinine analysis | 5 months

SECONDARY OUTCOMES:
Analyzing the differences in the measured concentrations in the dried blood spot made with blood obtained from venous sampling and capillary sampling. | 5 months
Evaluating the need of a correction factor and optimizing the correction factor when measuring the hematocrit in the DBS samples | 5 months
To investigate the patients' experience with the DBS method in comparison to venipuncture | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Brenda de Winter, PharmD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No